CLINICAL TRIAL: NCT07333755
Title: New Technique of End-to-Side Two-Layered Duct-to-Mucosa Pancreaticojejunostomy With Omental Wrapping and Glue (Glubran 2) During Laparoscopic Whipple Operation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mahmoud Rady, Lecturer of general surgery, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT (672)
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Periampullary Carcinoma Resectable
Keywords: pancreaticoduodenectomy; omental flaps; Laparoscopic whipple operation
MeSH Terms: interventions — Pancreaticojejunostomy; Adhesives

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A double-layered, end-to-side pancreaticojejunostomy without omental patch or glue (Active Comparator)
  Interventions: Procedure: Pancreaticojejunostomy without omental patch
- A double-layered, end-to-side pancreaticojejunostomy with omental patch and Glue (Active Comparator)
  Interventions: Procedure: Pancreaticojejunostomy with omental patch and glue

INTERVENTIONS:
Procedure: Pancreaticojejunostomy without omental patch — A laparoscopic pancreaticoduodenectomy with pylorus preservation was performed on each patient. A pancreatojejunostomy was created and not fixed with an omental patch or glue.
  Arms: A double-layered, end-to-side pancreaticojejunostomy without omental patch or glue
Procedure: Pancreaticojejunostomy with omental patch and glue — A laparoscopic pancreaticoduodenectomy was performed on each patient. A pancreaticojejunostomy was fixed with glue to secure the anastomosis. The greater omentum was separated longitudinally over an avascular zone, and one or two omental branches of the gastroepiploic arteries were preserved using pedicle omental flaps. The omentum was rolled up and secured with glue.
  Arms: A double-layered, end-to-side pancreaticojejunostomy with omental patch and Glue

SUMMARY:
Following pancreaticoduodenectomy, omental flaps around the pancreatic anastomosis and adhesive glue can lower the risk of pancreatic fistula, post-pancreatectomy bleeding, and delayed gastric emptying. The overall morbidity following pancreaticoduodenectomy can be decreased with this straightforward and efficient treatment.

ELIGIBILITY:
Inclusion Criteria:

- Resectable tumors of the periampullary region

Exclusion Criteria:

* Pancreatic or duodenal tumors
* Irresectability criteria (such as metastases, ascites, or arterial vascular invasion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
The rate of pancreatic fistula after pancreaticoduodenectomy | 4 weeks postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared upon request from the principle investigator.

REFERENCES:
- [Result] Maeda A, Ebata T, Kanemoto H, Matsunaga K, Bando E, Yamaguchi S, Uesaka K. Omental flap in pancreaticoduodenectomy for protection of splanchnic vessels. World J Surg. 2005 Sep;29(9):1122-6. doi: 10.1007/s00268-005-7900-3. PMID 16132400